CLINICAL TRIAL: NCT00744692
Title: A Pilot Study of Reduced Intensity Conditioning in Pediatric Patients <21 Years of Age With Non-Malignant Disorders Undergoing Umbilical Cord Blood Transplantation
Brief Title: Reduced Intensity Conditioning for Umbilical Cord Blood Transplant in Pediatric Patients With Non-Malignant Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008753
Record Dates: First submitted 2008-08-28; First posted 2008-09-01 (Estimated); Results first posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-07

CONDITIONS: Non Malignant Disorders; Immunodeficiencies; Congenital Marrow Failures; Hemoglobinopathies; Inborn Errors of Metabolism; Sickle Cell; Thalassemia; Lysosomal Storage Disease
Keywords: Immunodeficiencies; Congenital Marrow Failures; Hemoglobinopathies; Inborn Errors of Metabolism; SCIDS; Wiskott Aldrich; FEL; HLH; IPEX; LAD; Sickle Cell; Thalassemia; Omenn's Syndrome; Hurler's Syndrome; MLD; ALD; Sanfilippo; Krabbe; Hunter's syndrome; TaySachs; Diamond Blackfan Anemia; transplant; MPS; Gaucher
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Hemoglobinopathies; Metabolism, Inborn Errors; Thalassemia; Lysosomal Storage Diseases; Severe Combined Immunodeficiency; Mucopolysaccharidosis I; Mucopolysaccharidosis II; Anemia, Diamond-Blackfan | interventions — Alemtuzumab; Hydroxyurea; fludarabine; Melphalan; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RIC Cord Blood Transplant (Experimental): Reduced Intensity Conditioning for Umbilical Cord Blood Transplant
  Interventions: Biological: Unrelated Umbilical Cord Blood Transplant; Drug: Reduced Intensity Conditioning

INTERVENTIONS:
Biological: Unrelated Umbilical Cord Blood Transplant — Reduced Intensity Conditioning for unrelated umbilical cord blood transplant
Drug: Reduced Intensity Conditioning
  Other Names: Campath; Hydroxyurea; Fludarabine; Melphalan; Thiotepa

SUMMARY:
The primary objective is to determine the feasibility of attaining acceptable rates of donor cell engraftment (>25% donor chimerism at 180 days) following reduced intensity conditioning (RIC) regimens in pediatric patients < 21 years receiving cord blood transplantation for non-malignant disorders.

DETAILED DESCRIPTION:
Myeloablative doses of chemotherapy and/or radiation therapy are employed with the primary purpose of eradicating malignant cells. Additionally, these regimens exert varying degree of immunosuppression/immunoablation that aids in reducing the likelihood of rejection by host hematopoietic cells. However, myeloablative /immunoablative regimens have also been associated with significant regimen related toxicity (RRT) and regimen related mortality (RRM) that may cause death in up to 20% of patients and significantly higher rate of severe organ dysfunction or failure. While most of these RRT occur typically in the first 100 days [ e.g. VOD (veno occlusive disease), pulmonary or intracranial hemorrhage, multiorgan failure (MOF)], there are significant long term toxicities of TBI and/or chemotherapy including growth impairment, gonadal dysfunction/failure, hypothyroidism, cataracts, neurocognitive impairment, and second malignancies.

The primary objective is to determine the feasibility of attaining acceptable rates of donor cell engraftment (>25% donor chimerism at 180 days) following reduced intensity conditioning (RIC) regimens in pediatric patients < 21 years receiving cord blood transplantation for non-malignant disorders.

The secondary objectives are:

* To describe the pace of neutrophil and platelet recovery
* To evaluate the pace of immune reconstitution.
* To determine the treatment related mortality, overall survival and disease free survival by days 100 and 180 post-transplant
* To describe incidence of acute Graft Versus Host Disease (GVHD) (II - IV) and chronic extensive GVHD
* To describe the incidence of grade 3-4 organ toxicity
* To evaluate long-term complications, such as sterility, endocrinopathy, and growth failure
* To evaluate the incidence of late graft failures at 2 years post-transplant

ELIGIBILITY:
Inclusion Criteria:

* 0-21 years of age with a diagnosis of a immunodeficiency, congenital marrow failure syndrome, inborn error of metabolism, or hereditary anemia
* Appropriately matched related or unrelated umbilical cord blood unit with a cell dose ≥ 3 x 10e7cells/kg
* Performance score (lansky or karnofsky) greater than or equal to 70
* Adequate organ function (Creatinine ≤ 2.0 mg/dl and creatinine clearance ≥ 50 ml/min/1.73 m2; Hepatic transaminases (ALT/AST) ≤ 4 x normal; Shortening fraction >26% or ejection fraction >40% or > 80% of normal value for age; Pulmonary function tests demonstrating CVC or FEV1/FVC of >60% of predicted for age.)
* Informed consent
* Not pregnant or breast feeding
* Minimum life expectancy of at least 6 months
* HIV negative
* No uncontrolled infections at the time of cytoreduction
* Disease specific inclusion criteria

Exclusion Criteria:

* Patients with hemoglobinopathies > 3 years of age
* UCB unit with a total nucleated cell count < 3 x 10e7/kg or > 2 antigen mismatching
* Available HLA-matched related living donor able to donate without previous UCB donation
* Allogeneic hematopoietic stem cell transplant within the previous 6 months
* Any active malignancy, MDS, or any history of malignancy
* Severe acquired aplastic anemia
* DLCO < 60% of normal value for age; requirement for supplemental oxygen
* Uncontrolled bacterial, viral or fungal infection (currently taking medication and progression of clinical symptoms)
* Pregnancy or nursing mother
* HIV/HTLV seropositive, Hep B surface antigen positive, or HCV RNA positive by PCR
* Any condition that precludes serial follow-up

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2008-10; Primary Completion 2012-12 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suhag Parikh, MD, Principal Investigator — Duke Pediatric Blood and Marrow Transplant
Locations (1):
- Duke University Medical Center Pediatric Blood and Marrow Transplant Program, Durham, North Carolina, United States

REFERENCES:
- [Derived] Parikh SH, Mendizabal A, Benjamin CL, Komanduri KV, Antony J, Petrovic A, Hale G, Driscoll TA, Martin PL, Page KM, Flickinger K, Moffet J, Niedzwiecki D, Kurtzberg J, Szabolcs P. A novel reduced-intensity conditioning regimen for unrelated umbilical cord blood transplantation in children with nonmalignant diseases. Biol Blood Marrow Transplant. 2014 Mar;20(3):326-36. doi: 10.1016/j.bbmt.2013.11.021. Epub 2013 Dec 1. PMID 24296492

RESULTS

PARTICIPANT FLOW:
Groups:
- RIC Cord Blood Transplant: Reduced Intensity Conditioning for Umbilical Cord Blood Transplant
  Unrelated Umbilical Cord Blood Transplant: Reduced Intensity Conditioning for unrelated umbilical cord blood transplant
  Reduced Intensity Conditioning
Period: Overall Study
Arm/Group | RIC Cord Blood Transplant
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 22 subjects undergoing umbilical cord blood transplant
Arm/Group | RIC Cord Blood Transplant
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] — Age (in years) on the day of transplant
  years | 2.83 [0.3 to 8]
Age, Categorical [Count of Participants; unit: Participants] — Age (years) on the day of transplant
  Participants
    <=18 years | 22
    Between 18 and 65 years | 0
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Determine the Feasibility of Attaining Acceptable Rates of Donor Cell Engraftment (>25% Donor Cells at 180 Days) Following RIC Regimens in Children < 21 Years Receiving UCBT for Non-malignant Disorders.
Description: Determine the feasibility of attaining acceptable rates of donor cell engraftment (>25% donor cells at 180 days) following reduced intensity conditioning regimens in children < 21 years receiving cord blood transplant for non-malignant disorders.
Time Frame: 180 days post transplant
Population: Of the 22 patients enrolled, 18 patients were alive at 180 days, the time-point for primary end point
Measure: Number; unit: % of participants
Arm/Group | RIC Cord Blood Transplant
Number analyzed (Participants) | 18
% of participants | 88

2. Secondary Outcome: To Describe the Pace of Neutrophil Recovery
Description: Neutrophil recovery was defined as the first day of an absolute neutrophil count (ANC) more than 500/uL for 3 consecutive days not secondary to granulocyte infusions
Time Frame: 42 days post transplant
Measure: Median (Full Range); unit: days
Arm/Group | RIC Cord Blood Transplant
Number analyzed (Participants) | 22
days | 20 [12 to 28]

3. Secondary Outcome: To Evaluate the Pace of Immune Reconstitution.
Description: Immune reconstitution after RIC in UCBT was described. CD4 count is a standard measure of immune reconstitution and is described here. Additional data is available upon request.
Time Frame: 1 year post transplant
Population: Of the 22 patients at baseline, 5 patients died early before a year; and 2 additional patients had early graft failure. Thus 7 patients were not available for analysis of Immune reconstitution endpoint. CD4 count is reported here.
Measure: Median (Full Range); unit: cells/uL
Arm/Group | RIC Cord Blood Transplant
Number analyzed (Participants) | 15
cells/uL | 805 [6 to 2013]

4. Secondary Outcome: To Determine the Overall Survival at day180 Post-transplant
Description: To determine the overall survival at day180 post-transplant: determined by Kaplan Meier survival analysis
Time Frame: 180 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RIC Cord Blood Transplant
Number analyzed (Participants) | 22
percentage of participants | 81.8 [58.5 to 92.8]

5. Secondary Outcome: To Describe Incidence of Acute Graft Versus Host Disease (GVHD) (II - IV)
Description: To describe incidence of acute Graft Versus Host Disease (GVHD) (II - IV) : measured by cumulative incidence analysis
Time Frame: 100 days post transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RIC Cord Blood Transplant
Number analyzed (Participants) | 22
percentage of participants | 22.7 [5.3 to 40.1]

6. Secondary Outcome: To Describe the Incidence of Grade 3-4 Organ Toxicity
Time Frame: 2 years post transplant
Measure: Number; unit: participants
Arm/Group | RIC Cord Blood Transplant
Number analyzed (Participants) | 22
participants | 0

7. Secondary Outcome: To Evaluate Long-term Complications, Such as Sterility, Endocrinopathy, and Growth Failure
Time Frame: at least 2 years post transplant
Population: Of the 22 patients at baseline, 5 patients died early before a year; and 2 additional patients had early graft failure. Thus 7 patients were not available for analysis of this 2 year late effects endpoint.
Measure: Number; unit: percentage of patients
Arm/Group | RIC Cord Blood Transplant
Number analyzed (Participants) | 15
percentage of patients | 0

8. Secondary Outcome: To Evaluate the Incidence of Late Graft Failures at 2 Years Post-transplant
Time Frame: 2 years post transplant
Population: Of the 22 patients at baseline, 5 patients died early before a year; and 2 additional patients had early graft failure. Thus 7 patients were not available for analysis of this 2 year late graft failure endpoint.
Measure: Number; unit: participants
Arm/Group | RIC Cord Blood Transplant
Number analyzed (Participants) | 15
participants | 0

9. Secondary Outcome: To Describe the Pace of Platelet Recovery
Description: Platelet engraftment was defined as the first day of platelet counts more than 50,000/uL for 7 consecutive days without transfusions
Time Frame: 180 days post transplant
Measure: Median (Full Range); unit: days
Arm/Group | RIC Cord Blood Transplant
Number analyzed (Participants) | 22
days | 48 [33 to 144]

ADVERSE EVENTS:
Description: Adverse events that were expected and non-serious were not collected in this study.
Arm/Group | RIC Cord Blood Transplant
Serious Adverse Events (participants affected / at risk) | 18/22
Other Adverse Events (participants affected / at risk) | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RIC Cord Blood Transplant (N=22)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2
Fever (Investigations) | 5
Dehydration (Metabolism and nutrition disorders) | 2
Auto Immune Hemolytic Anemia (Blood and lymphatic system disorders) | 2
Infection (Infections and infestations) | 12
Hemolytic Transfusion Reaction (Blood and lymphatic system disorders) | 1
Graft Failure Post Transplant (Blood and lymphatic system disorders) | 2
Sepsis (Infections and infestations) | 3
Abdominal Pain (Gastrointestinal disorders) | 1
Nephrotic Syndrome (Renal and urinary disorders) | 1
VP Shunt Malfunction (Nervous system disorders) | 1
GI Distress (Gastrointestinal disorders) | 3
Multi System Organ Failure (General disorders) | 2
Seizure (Nervous system disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Graft Versus Host Disease (General disorders) | 4
Central Line Removal (Surgical and medical procedures) | 1
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 1
Hyperglycemia (Endocrine disorders) | 1
Pnematosis (Gastrointestinal disorders) | 1
Posterior Reversible Encephalopathy Syndrome (Nervous system disorders) | 1
Necrotic Ulcer (skin) (Skin and subcutaneous tissue disorders) | 1
Dental Rehabilitation (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes